CLINICAL TRIAL: NCT00762034
Title: Randomized, Open-Label, Phase 3 Study of Pemetrexed Plus Carboplatin and Bevacizumab Followed by Maintenance Pemetrexed and Bevacizumab Versus Paclitaxel Plus Carboplatin and Bevacizumab Followed by Maintenance Bevacizumab in Patients With Stage IIIB or IV Nonsquamous Non-Small Cell Lung Cancer
Brief Title: A Study of Pemetrexed, Carboplatin and Bevacizumab in Participants With Nonsquamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9707; H3E-MC-JMHD (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pem/Carbo/Bev (Experimental): Pemetrexed (Pem), carboplatin (Carbo) and bevacizumab (Bev) followed by pemetrexed and bevacizumab
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Biological: Bevacizumab
- Pac/Carbo/Bev (Active Comparator): Paclitaxel (Pac), carboplatin (Carbo) and bevacizumab (Bev) followed by bevacizumab
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — Induction therapy 500 milligram per meter squared (mg/m^2) intravenously (IV) every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days
  Other Names: Alimta; LY231514
  Arms: Pem/Carbo/Bev
Drug: Pemetrexed — Maintenance therapy 500 mg/m^2 IV every 21 days (with bevacizumab) until progressive disease or treatment discontinuation
  Other Names: Alimta; LY231514
  Arms: Pem/Carbo/Bev
Drug: Paclitaxel — Induction therapy 200 mg/m^2 IV every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days
  Arms: Pac/Carbo/Bev
Drug: Carboplatin — Induction therapy area under the concentration curve (AUC) 6 IV every 21 days for up to 4 cycles of 21 days
Biological: Bevacizumab — Induction therapy 15 milligrams per kilogram (mg/kg) IV every 21 days for up to 4 cycles of 21 days
Biological: Bevacizumab — Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.

SUMMARY:
This study will compare overall survival in participants with Stage IIIB or IV nonsquamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* You must sign an informed consent document for clinical research.
* You must have Stage IIIB or Stage IV nonsquamous non-small cell lung cancer.
* You must not have received any prior treatment for your disease.
* Prior radiation therapy is allowed to < 25% of the bone marrow; however, prior radiation to the whole pelvis is not allowed. If you have had radiation therapy to the chest, you are not eligible to participate.
* You must be at least 18 years of age or older.
* You must have measureable tumor lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) or disease can be evaluated on computed tomography (CT) scan.
* Your test results assessing the function of blood forming tissue, kidneys and liver must be satisfactory.
* Women must be sterile, postmenopausal or on contraception and men must be sterile (for example post-vasectomy) or on contraception.

Exclusion Criteria:

* You cannot have clinically significant third-space fluid collections (e.g. ascites or pleural effusions that cannot be controlled by drainage or other procedures).
* You cannot have Non-small Cell Lung Carcinoma (NSCLC) of predominantly squamous cell histology.
* You cannot have known central nervous system (CNS) disease, other than stable, treated brain metastasis.
* You cannot have undergone a surgical procedure, open biopsy, open pleurodesis, or significant traumatic injury within 28 days of starting the study treatment, or have an anticipated need for major surgery during the study.
* You cannot have a history of gastrointestinal fistula, perforation, or abscess, inflammatory bowel disease, or diverticulitis.
* You are currently receiving ongoing treatment with full-dose warfarin or equivalent.
* You cannot have significant vascular disease, serious cardiac conditions (such as heart attack), stroke or transient ischemic attack within 6 months of the trial.
* You cannot have evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
* You cannot have inadequately controlled hypertension, or a history of hypertensive crisis or hypertensive encephalopathy.
* You cannot have a serious, nonhealing wound, active ulcer, or untreated bone fracture.
* You cannot have another form of cancer, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within the last 5 years.
* You cannot have received an investigational treatment within 30 days prior to the trial.
* You cannot have previously received treatment with paclitaxel, carboplatin, pemetrexed, or bevacizumab.
* You cannot be pregnant or breast-feeding.
* You cannot have a known sensitivity to any component of paclitaxel, carboplatin, pemetrexed, or bevacizumab.
* You cannot have a history of hemoptysis (coughing blood) within 3 months prior to the trial.
* You are unable to stop taking aspirin more than 1.3 grams per day or other nonsteroidal anti-inflammatory drugs (NSAIDs).
* You are unable or unwilling to take folic acid or vitamin B12 supplementation.
* You are unable to take corticosteroids.
* You have any other on-going illnesses including active infections that may not allow you to adhere to the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2008-12; Primary Completion 2012-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMC - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (67):
- United States (67):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jonesboro, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alhambra, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bakersfield, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duarte, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fountain Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Verne, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rancho Mirage, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redondo Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Rosa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Junction, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Worth, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Saint Lucie, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuart, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Gordon, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gurnee, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Skokie, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Albany, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chevy Chase, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frederick, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Framingham, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lambertville, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duluth, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stony Brook, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kittanning, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willow Grove, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abingdon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin

REFERENCES:
- [Derived] Spigel DR, Patel JD, Reynolds CH, Garon EB, Hermann RC, Govindan R, Olsen MR, Winfree KB, Chen J, Liu J, Guba SC, Socinski MA, Bonomi P. Quality of life analyses from the randomized, open-label, phase III PointBreak study of pemetrexed-carboplatin-bevacizumab followed by maintenance pemetrexed-bevacizumab versus paclitaxel-carboplatin-bevacizumab followed by maintenance bevacizumab in patients with stage IIIB or IV nonsquamous non-small-cell lung cancer. J Thorac Oncol. 2015 Feb;10(2):353-9. doi: 10.1097/JTO.0000000000000277. PMID 25611228
- [Derived] Reynolds CH, Patel JD, Garon EB, Olsen MR, Bonomi P, Govindan R, Pennella EJ, Liu J, Guba SC, Li S, Spigel DR, Hermann RC, Socinski MA, Obasaju CK. Exploratory Subset Analysis of African Americans From the PointBreak Study: Pemetrexed-Carboplatin-Bevacizumab Followed by Maintenance Pemetrexed-Bevacizumab Versus Paclitaxel-Carboplatin-Bevacizumab Followed by Maintenance Bevacizumab in Patients With Stage IIIB/IV Nonsquamous Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2015 May;16(3):200-8. doi: 10.1016/j.cllc.2014.11.004. Epub 2014 Nov 18. PMID 25516338
- [Derived] Patel JD, Socinski MA, Garon EB, Reynolds CH, Spigel DR, Olsen MR, Hermann RC, Jotte RM, Beck T, Richards DA, Guba SC, Liu J, Frimodt-Moller B, John WJ, Obasaju CK, Pennella EJ, Bonomi P, Govindan R. PointBreak: a randomized phase III study of pemetrexed plus carboplatin and bevacizumab followed by maintenance pemetrexed and bevacizumab versus paclitaxel plus carboplatin and bevacizumab followed by maintenance bevacizumab in patients with stage IIIB or IV nonsquamous non-small-cell lung cancer. J Clin Oncol. 2013 Dec 1;31(34):4349-57. doi: 10.1200/JCO.2012.47.9626. Epub 2013 Oct 21. PMID 24145346
- [Derived] Patel JD, Bonomi P, Socinski MA, Govindan R, Hong S, Obasaju C, Pennella EJ, Girvan AC, Guba SC. Treatment rationale and study design for the pointbreak study: a randomized, open-label phase III study of pemetrexed/carboplatin/bevacizumab followed by maintenance pemetrexed/bevacizumab versus paclitaxel/carboplatin/bevacizumab followed by maintenance bevacizumab in patients with stage IIIB or IV nonsquamous non-small-cell lung cancer. Clin Lung Cancer. 2009 Jul;10(4):252-6. doi: 10.3816/CLC.2009.n.035. PMID 19632943

RESULTS

PARTICIPANT FLOW:
Groups:
- Pem/Carbo/Bev: Pemetrexed (Pem), carboplatin (Carbo) and bevacizumab (Bev) followed by pemetrexed and bevacizumab
  Bevacizumab: Induction therapy 15 milligrams per kilogram (mg/kg) intravenously (IV) every 21 days for up to 4 cycles of 21 days
  Bevacizumab: Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.
  Pemetrexed: Induction therapy 500 milligram per meter squared (mg/m^2) IV every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days
  Pemetrexed: Maintenance therapy 500 mg/m^2 IV every 21 days (with bevacizumab) until progressive disease or treatment discontinuation
  Carboplatin: Induction therapy of 6 area under the concentration curve (AUC 6) IV every 21 days for up to 4 cycles of 21 days
- Pac/Carbo/Bev: Paclitaxel (Pac), carboplatin (Carbo) and bevacizumab (Bev) followed by bevacizumab
  Paclitaxel: Induction therapy 200 milligram per meter squared (mg/m^2) intravenously (IV) every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days
  Bevacizumab: Induction therapy 15 mg/kg IV every 21 days for up to 4 cycles of 21 days
  Bevacizumab: Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.
  Carboplatin: Induction therapy 6 area under the concentration curve (AUC 6) IV every 21 days for up to 4 cycles of 21 days
Period: Induction Period
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Started | 472 | 467
Received at Least 1 Dose of Study Drug | 442 | 443
Completed | 294 | 298
Not Completed | 178 | 169
Not completed — Protocol Violation | 1 | 2
Not completed — Entry Criterion Not Met | 12 | 11
Not completed — Adverse Event | 27 | 38
Not completed — Lost to Follow-up | 1 | 1
Not completed — Progressive Disease | 73 | 55
Not completed — Physician Decision | 21 | 20
Not completed — Withdrawal by Subject | 15 | 19
Not completed — Deaths Not Due to Study Disease | 19 | 14
Not completed — Deaths Due to Study Disease | 9 | 9
Period: Maintenance Period
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Started | 294 | 298
Received at Least 1 Dose of Study Drug | 294 | 298
Completed | 0 | 0
Not Completed | 294 | 298
Not completed — Protocol Violation | 1 | 3
Not completed — Entry Criterion Not Met | 0 | 2
Not completed — Adverse Event | 42 | 26
Not completed — Progressive Disease | 186 | 224
Not completed — Physician Decision | 25 | 20
Not completed — Withdrawal by Subject | 34 | 14
Not completed — Death not due to study disease | 2 | 5
Not completed — Death due to study disease | 3 | 3
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev | Total
Number analyzed (Participants) | 472 | 467 | 939
Age, Customized [Number; unit: participants]
  <=65 years | 249 | 236 | 485
  >65 years | 223 | 231 | 454
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 218 | 439
  Male | 251 | 249 | 500
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 409 | 396 | 805
  Black or African American | 42 | 52 | 94
  Asian | 15 | 14 | 29
  American Indian or Alaska Native | 1 | 1 | 2
  Multiple race/ethnicities | 2 | 3 | 5
  Information not provided | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 472 | 467 | 939
Previously Treated Brain Metastasis [Number; unit: participants]
  Yes | 52 | 52 | 104
  No | 420 | 415 | 835
Histological Subtype [Number; unit: participants] — Non-small Cell Lung Carcinoma (NSCLC)
  participants
    Adenocarcinoma, Lung | 367 | 360 | 727
    Bronchioalveolar Carcinoma | 4 | 3 | 7
    Large Cell Lung Carcinoma | 8 | 15 | 23
    NSCLC Not Otherwise Specified | 47 | 39 | 86
    NSCLC Poorly Differentiated | 39 | 47 | 86
    Predominantly Adenocarcinoma | 7 | 2 | 9
    Unknown | 0 | 1 | 1
Histological Category for Subgroup Analyses [Number; unit: participants]
  Adenocarcinoma | 378 | 365 | 743
  Large Cell Carcinoma | 8 | 15 | 23
  Other or Indeterminant | 86 | 86 | 172
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) is the duration from date of randomization to date of death from any cause. Participants were censored at the date they were last known to be alive.
Time Frame: Baseline to date of death from any cause (up to 37.06 months)
Population: All randomized participants using the intent-to-treat principle. Number of participants censored: n=131, 127 in Pem/Carbo/Bev and Pac/Carbo/Bev arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
months | 12.55 [11.30 to 14.03] | 13.40 [11.86 to 14.91]
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.94896, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.86 to 1.16]

2. Secondary Outcome: Percentage of Participants With a Complete Response (CR) and Partial Response (PR) (Overall Response Rate)
Description: Overall Response Rate (ORR) is the number of participants with a Complete Response (CR) and Partial Response (PR) divided by the total number of randomized participants per arm, then multiplied by 100. Response is based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.0) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions compared to baseline or the complete disappearance of target lesions, with persistence of 1 or more nontarget lesion(s) and no new lesions.
Time Frame: Baseline to measured progressive disease (up to 37.06 months)
Population: All randomized participants using the intent-to-treat principle
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
percentage of participants | 34.1 [29.8 to 38.6] | 33.0 [28.7 to 37.4]
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.72997, Fisher Exact

3. Secondary Outcome: Percentage of Participants With a Complete Response (CR), Partial Response (PR), and Stable Disease (SD) (Disease Control Rate)
Description: Disease Control Rate (DCR) is the number of participants with a Complete Response (CR), Partial Response (PR), and Stable Disease (SD) divided by the total number of randomized participants per arm, then multiplied by 100. Response is based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.0) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions compared with baseline or the complete disappearance of target lesions, with persistence of 1 or more nontarget lesion(s) and no new lesions. Progressive Disease (PD) was defined as at least 20% increase in sum of longest diameter of target lesions compared with the smallest sum of the longest diameter recorded since the start of treatment or the appearance of 1 or more new lesion(s). Stable Disease (SD) was defined as small changes that did not meet above criteria.
Time Frame: Baseline to measured progressive disease (up to 37.06 months)
Population: All randomized participants using the intent-to-treat principle
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
percentage of participants | 65.9 [61.4 to 70.2] | 69.8 [65.4 to 73.9]
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.20892, Fisher Exact

4. Secondary Outcome: Progression Free Survival Time
Description: Progression free survival (PFS) is defined as the time from date of randomization to the date of objective disease progression or death due to any cause. Participants were censored at date of last PFS assessment prior to the cutoff date or the date of initiation of subsequent systemic anticancer therapy, whichever was earlier.
Time Frame: Baseline to measured progressive disease or date of death from any cause (up to 33.54 months)
Population: All randomized participants using the intent-to-treat principle. Number of participants censored: n=127, 109 in Pem/Carbo/Bev and Pac/Carbo/Bev arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
months | 6.04 [5.55 to 6.87] | 5.55 [5.39 to 5.98]
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.01206, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.71 to 0.96]

5. Secondary Outcome: Time to Progressive Disease
Description: Time to progressive disease was defined as the time from randomization to the first date of objective disease progression. Participants were censored at date of last PFS assessment prior to the cutoff date or the date of initiation of subsequent systemic anticancer therapy, whichever was earlier.
Time Frame: Baseline to measured progressive disease (up to 37.06 months)
Population: All randomized participants using the intent-to-treat principle. Number of participants censored: n=198, 172 in Pem/Carbo/Bev and Pac/Carbo/Bev arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
months | 7.03 [6.24 to 8.05] | 6.04 [5.58 to 6.87]
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.006, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.67 to 0.94]

6. Secondary Outcome: Safety and Toxicity Profile of Study Treatments
Description: Safety and toxicity profile was defined as serious and other non-serious adverse events. A summary of serious and all other non-serious adverse events is located in the Reported Adverse Event module.
Time Frame: Baseline to study endpoint (up to 37.06 months)
Population: All randomized participants who received at least 1 dose of study drug during the specified treatment phase.
Measure: Number; unit: participants
Groups:
- Pem/Carbo/Bev; Induction Phase; Pem/Carbo/Bev; Maintenance Phase: Pemetrexed (Pem), carboplatin (Carbo) and bevacizumab (Bev) followed by pemetrexed and bevacizumab
  Bevacizumab: Induction therapy 15 milligrams per kilogram (mg/kg) intravenously (IV) every 21 days for up to 4 cycles of 21 days
  Bevacizumab: Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.
  Pemetrexed: Induction therapy 500 milligram per meter squared (mg/m^2) IV every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days
  Pemetrexed: Maintenance therapy 500 mg/m^2 IV every 21 days (with bevacizumab) until progressive disease or treatment discontinuation
  Carboplatin: Induction therapy of 6 area under the concentration curve (AUC 6) IV every 21 days for up to 4 cycles of 21 days
- Pac/Carbo/Bev; Induction Phase; Pac/Carbo/Bev; Maintenance Phase: Paclitaxel (Pac), carboplatin (Carbo) and bevacizumab (Bev) followed by bevacizumab
  Paclitaxel: Induction therapy 200 milligram per meter squared (mg/m^2) intravenously (IV) every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days
  Bevacizumab: Induction therapy 15 mg/kg IV every 21 days for up to 4 cycles of 21 days
  Bevacizumab: Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.
  Carboplatin: Induction therapy 6 area under the concentration curve (AUC 6) IV every 21 days for up to 4 cycles of 21 days
Arm/Group | Pem/Carbo/Bev; Induction Phase | Pem/Carbo/Bev; Maintenance Phase | Pac/Carbo/Bev; Induction Phase | Pac/Carbo/Bev; Maintenance Phase
Number analyzed (Participants) | 442 | 292 | 443 | 298
participants
  Serious Adverse Events (SAEs) | 111 | 83 | 123 | 68
  Other Adverse Events (AEs) | 432 | 288 | 431 | 296

7. Secondary Outcome: Duration of Hospitalizations Per Participant
Description: Length of hospitalization in participants hospitalized during the study or within 30 days of discontinuation regardless of whether the hospitalization was or was not due to study drug.
Time Frame: Baseline to study endpoint (up to 37.06 months)
Population: All randomized participants who received at least 1 dose of study drug and had at least one hospitalization while on study or within 30 days of discontinuation.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 177 | 172
days | 9.4 (9.8) | 8.0 (6.7)

8. Secondary Outcome: Number of Participants Who Received a Transfusion
Time Frame: Baseline to study endpoint (up to 37.06 months)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 442 | 443
participants | 116 | 44

9. Secondary Outcome: Number of Participants Receiving Concomitant Medication
Time Frame: Baseline to study endpoint (up to 37.06 months)
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
participants | 406 | 421

10. Secondary Outcome: Change From Baseline in Participant Reported Outcomes as Assessed by the Functional Assessment of Cancer Therapy - General (FACT-G)
Description: The FACT-G is a validated instrument used to measure quality of life (QOL) in participants with cancer consisting of the 27-item questionnaire and is organized into subscales, each designed to assess a QOL domain: physical well-being (PWB)-7 items; social/family well-being (SWB)-7 items; emotional well-being (EWB)-6 items; functional well-being (FWB)-7 items. Each item uses a 5 point rating scale (0="not at all" and 4=equals "very much"). FACT-G Total is the sum of the scores of all 4 subscales and ranges from 0 to 108. Higher scores indicate better QOL. Least squares mean (LSmean) change is calculated using the linear-mixed model (LMM) analysis controlled for treatment, baseline value, time point and treatment by time point interaction.
Time Frame: Baseline, up to first 10 cycles (4 induction and 6 maintenance cycles, cycle=21 days)
Population: The LMM analysis includes data from all participants in each arm for whom a validated translation is available in a language in which the completer (participant) is fluent and have evaluable FACT-G data, using the intent-to-treat principle.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 462
units on a scale | 0.51 (0.54) | 0.18 (0.54)
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.667, Mixed Models Analysis — Mixed Model Analysis has treatment, baseline, time point, and treatment by timepoint interaction as fixed effects

11. Secondary Outcome: Change From Baseline in Participant Reported Outcomes as Assessed by the Functional Assessment of Cancer Therapy - Lung (FACT-L)
Description: FACT-L is a valid instrument used to measure quality of life (QOL) in participants with cancer consisting of the 27-item FACT-General (G) and 9-item lung cancer subscale (LCS). FACT-G is organized into subscales: physical well-being (PWB)-7 items; social/family well-being (SWB)-7 items; emotional well-being (EWB)-6 items; functional well-being (FWB)-7 items. Each item uses a 5 point rating scale (0="not at all" and 4=equals "very much"). FACT-L Total Score=4 subscales + LCS and ranges from 0 to 144. Trial Outcome Index-Lung (TOI-L)=PWB+FWB+LCS and ranges from 0 to 92. Higher scores indicate better QOL. Least squares mean (LSmean) change is calculated using the linear-mixed model (LMM) analysis controlled for treatment, baseline value, time point and treatment by time point interaction.
Time Frame: Baseline, up to first 10 cycles (4 induction and 6 maintenance cycles, cycle=21 days)
Population: The LMM analysis includes data from all participants in each arm for whom a validated translation is available in a language in which the completer (participant) is fluent and have evaluable FACT-L, using the intent-to-treat principle.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
units on a scale
  FACT-L Total Score (n=397, 392) | 1.88 (0.65) | 1.66 (0.66)
  Trial Outcome Index-Lung (TOI-L) (n=396, 394) | -0.38 (0.50) | -0.40 (0.50)
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.815, Mixed Models Analysis — p-value for FACT-L Total; Mixed Model Analysis has treatment, baseline, time point, and treatment by timepoint interaction as fixed effects
Statistical Analysis 2: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.978, Mixed Models Analysis — p-value for FACT-L TOI; Mixed Model Analysis has treatment, baseline, time point, and treatment by timepoint interaction as fixed effects

12. Secondary Outcome: Change From Baseline in Participant Reported Outcomes as Assessed by the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group- Neurotoxicity (FACT/GOG-Ntx)
Description: FACT/GOG-Ntx is a validated instrument used to measure quality of life (QOL) in participants with cancer and neurotoxicity (Ntx) consisting of 27-item FACT-General (G) and 11-item Ntx subscale. FACT-G is organized into domain subscales: physical well-being (PWB)-7 items; social/family well-being (SWB)-7 items; emotional well-being (EWB)-6 items; functional well-being (FWB)-7 items; each uses a 5 point rating scale (0="not at all" and 4=equals "very much"). FACT/GOG-Ntx Total Score=sum 5 subscales and ranges from 0-152. Ntx Trial Outcome Index (TOI-Ntx)=PWB+FWB+NTX and range from 0-100. For all FACT scales, higher scores indicate better QOL. Least squares mean (LSmean) change is calculated using the linear-mixed model (LMM) analysis controlled for treatment, baseline value, time point and treatment by time point interaction.
Time Frame: Baseline, up to first 10 cycles (4 induction and 6 maintenance cycles, cycle=21 days)
Population: The LMM analysis includes data from all participants in each arm for whom a validated translation is available in a language in which the completer (participant) is fluent and have evaluable FACT/GOG-Ntx data, using the intent-to-treat principle.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 472 | 467
units on a scale
  FACT/GOG-Ntx Total Score (n=393, 389) | -0.60 (0.70) | -5.48 (0.70)
  Ntx Trial Outcome Index (TOI-Ntx)(n=393, 390) | -2.79 (0.55) | -7.60 (0.55)
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value for FACT/GOG-Ntx Total; Mixed Model Analysis has treatment, baseline, time point, and treatment by timepoint interaction as fixed effects
Statistical Analysis 2: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value for FACT/GOG-Ntx TOI; Mixed Model Analysis has treatment, baseline, time point, and treatment by timepoint interaction as fixed effects

13. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) for Pemetrexed
Time Frame: Cycle 1 (pre-dose, 0.17, 0.33, 0.58, 0.83, 1, 1.75, 2.5, 4. 6. 8, and 24 hours post-dose)
Population: Participants who were randomized to Pem/Carbo/Bev, who received study drug, and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Groups:
- Pem/Carbo/Bev: Pemetrexed (Pem), carboplatin (Carbo) and bevacizumab (Bev)followed by pemetrexed and bevacizumab
  Bevacizumab: Induction therapy 15 milligrams per kilogram (mg/kg) intravenously (IV) every 21 days for up to 4 cycles of 21 days
  Bevacizumab: Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.
  Pemetrexed: Induction therapy 500 milligram per meter squared (mg/m^2) IV every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days
  Pemetrexed: Maintenance therapy 500 mg/m^2 IV every 21 days (with bevacizumab) until progressive disease or treatment discontinuation
  Carboplatin: Induction therapy of 6 area under the concentration curve (AUC 6) IV every 21 days for up to 4 cycles of 21 days
Arm/Group | Pem/Carbo/Bev
Number analyzed (Participants) | 14
micrograms per milliliter (μg/mL) | 122 (20)

14. Secondary Outcome: Pharmacokinetics (PK): Elimination Half-life (t1/2) for Pemetrexed
Time Frame: Cycle 1 (pre-dose, 0.17, 0.33, 0.58, 0.83, 1, 1.75, 2.5, 4. 6. 8, and 24 hours post-dose)
Population: Participants who were randomized to Pem/Carbo/Bev, who received study drug, and had evaluable t1/2 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hr)
Arm/Group | Pem/Carbo/Bev
Number analyzed (Participants) | 15
hours (hr) | 2.88 (13)

15. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Zero to Infinity (AUC(0-∞)) for Pemetrexed
Time Frame: Cycle 1 (pre-dose, 0.17, 0.33, 0.58, 0.83, 1, 1.75, 2.5, 4. 6. 8, and 24 hours post-dose)
Population: Participants who were randomized to Pem/Carbo/Bev, who received study drug, and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg•hr/mL)
Arm/Group | Pem/Carbo/Bev
Number analyzed (Participants) | 15
microgram*hour per milliliter (μg•hr/mL) | 203 (23)

16. Secondary Outcome: Pharmacokinetics (PK): Pemetrexed Clearance (CL)
Time Frame: Cycle 1 (pre-dose, 0.17, 0.33, 0.58, 0.83, 1, 1.75, 2.5, 4. 6. 8, and 24 hours post-dose)
Population: Participants who were randomized to Pem/Carbo/Bev, who received study drug, and had evaluable CL data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per minute (mL/min)
Arm/Group | Pem/Carbo/Bev
Number analyzed (Participants) | 15
milliliters per minute (mL/min) | 72.1 (25)

17. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) for Total (Bound and Unbound) Platinum and Unbound Platinum
Description: Platinum is a metabolite of Carboplatin (Carbo) and is found in the blood as both a bound and unbound form.
Time Frame: Cycle 1 (pre-dose, 0.25, 0.5, 0.67, 1.42, 2.17, 4, 6, 8, 24, 48, and 72 hours post-dose)
Population: Randomized participants who received study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 20 | 16
micrograms per milliliter (μg/mL)
  Total (Bound and Unbound) | 18.4 (24) | 17.8 (33)
  Unbound (n=18, 15) | 21.1 (31) | 17.1 (34)

18. Secondary Outcome: Pharmacokinetics (PK): Elimination Half-life (t1/2) for Total (Bound and Unbound) Platinum and Unbound Platinum
Description: Platinum is a metabolite of Carboplatin (Carbo) and is found in the blood as both a bound and unbound form.
Time Frame: Cycle 1 (pre-dose, 0.25, 0.5, 0.67, 1.42, 2.17, 4, 6, 8, 24, 48, and 72 hours post-dose)
Population: Randomized participants who received study drug and had evaluable t1/2 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hr)
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 18 | 16
hours (hr)
  Total (Bound and Unbound) | 65.6 (69) | 86.4 (21)
  Unbound (n=17, 13) | 2.03 (15) | 1.95 (21)

19. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Zero to Infinity (AUC(0-∞)) for Total (Bound and Unbound) Platinum and Unbound Platinum
Description: Platinum is a metabolite of Carboplatin (Carbo) and is found in the blood as both a bound and unbound form.
Time Frame: Cycle 1 (pre-dose, 0.25, 0.5, 0.67, 1.42, 2.17, 4, 6, 8, 24, 48, and 72 hours post-dose)
Population: Randomized participants who received study drug and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg•hr/mL)
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 18 | 16
microgram*hour per milliliter (μg•hr/mL)
  Total (Bound and Unbound) | 160 (32) | 182 (24)
  Unbound (n=17, 13) | 55.7 (33) | 62.9 (34)

20. Secondary Outcome: Pharmacokinetics (PK): Platinum Clearance (CL) for Total (Bound and Unbound) and Unbound Forms
Description: Platinum is a metabolite of Carboplatin (Carbo) and is found in the blood as both a bound and unbound form.
Time Frame: Cycle 1 (pre-dose, 0.25, 0.5, 0.67, 1.42, 2.17, 4, 6, 8, 24, 48, and 72 hours post-dose)
Population: Randomized participants who received study drug and had evaluable CL data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 18 | 16
liters per hour (L/hr)
  Total (Bound and Unbound) | 2.02 (39) | 1.87 (28)
  Unbound (n=17, 13) | 5.81 (35) | 5.36 (47)

21. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) for Bevacizumab
Time Frame: Cycle 1 (pre-dose, 0.75, 1.5, 3, 5, 7, 24, 48, 72, 168, 336, and 503 hours post-dose)
Population: Randomized participants who received study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 20 | 16
micrograms per milliliter (μg/mL) | 276 (18) | 302 (20)

22. Secondary Outcome: Pharmacokinetics (PK): Elimination Half-life (t1/2) for Bevacizumab
Time Frame: Cycle 1 (pre-dose, 0.75, 1.5, 3, 5, 7, 24, 48, 72, 168, 336, and 503 hours post-dose)
Population: Randomized participants who received study drug and had evaluable t1/2 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 17 | 16
days | 14.8 (36) | 12.8 (46)

23. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Zero to Infinity (AUC(0-∞)) Bevacizumab
Time Frame: Cycle 1 (pre-dose, 0.75, 1.5, 3, 5, 7, 24, 48, 72, 168, 336, and 503 hours post-dose)
Population: Randomized participants who received study drug and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg•day/mL)
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 17 | 16
microgram*day per milliliter (μg•day/mL) | 3070 (29) | 3160 (33)

24. Secondary Outcome: Pharmacokinetics (PK): Bevacizumab Clearance (CL)
Time Frame: Cycle 1 (pre-dose, 0.75, 1.5, 3, 5, 7, 24, 48, 72, 168, 336, and 503 hours post-dose)
Population: Randomized participants who received study drug and had evaluable CL data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per day (L/day)
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 17 | 16
liters per day (L/day) | 0.341 (31) | 0.376 (38)

25. Secondary Outcome: Translational Research: Number of Participants With Epidermal Growth Factor Receptor (EGFR) Mutations
Description: Epidermal Growth Factor Receptor (EGFR) mutations were measured by polymerase chain reaction (PCR).
Time Frame: Baseline
Population: All randomized participants with EGFR data regardless of study treatment.
Measure: Number; unit: participants
Groups:
- Pem or Pac Plus Carbo/Bev: Participants who received either Pem/Carbo/Bev or Pac/Carbo/Bev treatment.
  Pem/Carbo/Bev Treatment-500 mg per meter squared (mg/m^2) Pem IV every 21 days, plus Carbo AUC 6 IV every 21 days for up to first 4 cycles of 21 days, plus 15 mg/kg Bev IV every 21.
  OR
  Pac/Carbo/Bev Treatment-200 mg/m^2 Pac IV and AUC 6 Carbo IV every 21 days for up to first 4 cycles of 21 days, plus 15 mg/kg Bev IV every 21 days.
Arm/Group | Pem or Pac Plus Carbo/Bev
Number analyzed (Participants) | 132
participants
  EGFR mutation positive | 11
  EGFR mutation negative | 121

26. Secondary Outcome: Translational Research: Overall Survival (OS) Based on Nuclear Thyroid Transcription Factor-1 (TTF-1) Expression Regardless of Study Treatment
Description: Nuclear Thyroid Transcription Factor-1 (TTF-1) expression was measured using an Immunohistochemistry (IHC) assay which were scored using a 0 (negative, no staining) to 3+ (brightest staining) scoring system, and H score is a calculated using formula: 1x(percentage of cells stained 1+) + 2x(percentage of cells stained 2+) + 3x(percentage of cells stained 3+). TTF-1 Positive have an H score >0 and TTF-1 Negative have an H score=0. Overall survival (OS) is the duration from date of randomization to date of death from any cause. Participants were censored at the date they were last known to be alive.
Time Frame: Baseline to date of death from any cause (up to 37.06 months)
Population: All randomized participants with TTF-1 H scores regardless of study treatment. Participants censored: n=38, 11 in the TTF-1 Nuclear Positive and Negative arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- TTF-1 Positive (H Score > 0): Participants who were TTF-1 Positive (H score > 0) and received either Pem/Carbo/Bev or Pac/Carbo/Bev treatment.
  Pem/Carbo/Bev Treatment-500 mg per meter squared (mg/m^2) Pem IV every 21 days, plus Carbo AUC 6 IV every 21 days for up to first 4 cycles of 21 days, plus 15 mg/kg Bev IV every 21.
  OR
  Pac/Carbo/Bev Treatment-200 mg/m^2 Pac IV and AUC 6 Carbo IV every 21 days for up to first 4 cycles of 21 days, plus 15 mg/kg Bev IV every 21 days.
- TTF-1 Negative (H Score = 0): Participants who were TTF-1 Negative (H score = 0) and received either Pem/Carbo/Bev or Pac/Carbo/Bev treatment.
  Pem/Carbo/Bev Treatment-500 mg per meter squared (mg/m^2) Pem IV every 21 days, plus Carbo AUC 6 IV every 21 days for up to first 4 cycles of 21 days, plus 15 mg/kg Bev IV every 21.
  OR
  Pac/Carbo/Bev Treatment-200 mg/m^2 Pac IV and AUC 6 Carbo IV every 21 days for up to first 4 cycles of 21 days, plus 15 mg/kg Bev IV every 21 days.
Arm/Group | TTF-1 Positive (H Score > 0) | TTF-1 Negative (H Score = 0)
Number analyzed (Participants) | 139 | 66
months | 14.9 [12.8 to 17.6] | 8.7 [6.4 to 10.5]
Statistical Analysis 1: Comparison: TTF-1 Positive (H Score > 0) vs TTF-1 Negative (H Score = 0); Test type: Superiority or Other; p < 0.001, Regression, Cox — p-value was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.480, 95% CI 2-sided [0.338 to 0.681]

27. Secondary Outcome: Translational Research: Overall Survival (OS) Based on Cytoplasmic and Nuclear Thymidylate Synthase (TS) Expression
Description: Cytoplasmic and nuclear Thymidylate Synthase (TS) expression was measured using an Immunohistochemistry (IHC) assay which were scored using a 0 (negative, no staining) to 3+ (brightest staining) scoring system for cytoplasmic and nuclear staining, and H score was calculated using formula: 1x(percentage of cells stained 1+) + 2x(percentage of cells stained 2+) + 3x(percentage of cells stained 3+). TS Positive have an H score >0 and TS Negative have an H score=0. Overall survival (OS) is the duration from date of randomization to date of death from any cause. Participants were censored at the date they were last known to be alive.
Time Frame: Baseline to date of death from any cause (up to 37.06 months)
Population: All randomized participants with TS Cytoplasm and Nucleus H scores. Participants censored: TS Cytoplasm Positive n=23, 20 and Negative n=4, 1; TS Nucleus Positive n=17, 9 and Negative n=10, 12 for the Pem/Carbo/Bev and Pac/Carbo/Bev arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 100 | 89
months
  TS Cytoplasm Positive (H score > 0; n=90, 83) | 12.9 [10.8 to 16.9] | 12.4 [10.9 to 15.5]
  TS Cytoplasm Negative (H score = 0; n=10, 6) | 18.2 [12.5 to NA] — Not calculable due to the low number of participants reaching endpoint event of death. | 11.6 [9.1 to 14.7]
  TS Nucleus Positive (H score > 0; n=68, 51) | 12.7 [9.7 to 15.4] | 12.4 [8.4 to 15.5]
  TS Nucleus Negative (H score = 0; n=32, 38) | 19.2 [12.5 to 24.1] | 12.4 [10.1 to 17.1]
Statistical Analysis 1: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.673, Regression, Cox — p-value is for TS Cytoplasm Positive (H score > 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.927, 95% CI 2-sided [0.654 to 1.316]
Statistical Analysis 2: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.287, Regression, Cox — p-value is for TS Cytoplasm Negative (H score = 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.521, 95% CI 2-sided [0.157 to 1.729]
Statistical Analysis 3: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.2, Regression, Cox — p-value is for TS Nucleus Positive (H score > 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.759, 95% CI 2-sided [0.498 to 1.157]
Statistical Analysis 4: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.915, Regression, Cox — p-value is for TS Nucleus Negative (H score = 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.969, 95% CI 2-sided [0.540 to 1.738]

28. Secondary Outcome: Translational Research: Overall Survival (OS) Based on Cytoplasmic and Membrane Folate Receptor Alpha (FR-α) Expression
Description: Cytoplasmic and membrane Folate Receptor Alpha (FR-α) expression was measured using an Immunohistochemistry (IHC) assay which were scored using a 0 (negative, no staining) to 3+ (brightest staining) scoring system for cytoplasmic or membrane staining, and H score is a calculated using formula: 1x(percentage of cells stained 1+) + 2x(percentage of cells stained 2+) + 3x(percentage of cells stained 3+). FR-α Positive have an H score >0 and FR-α Negative have an H score=0. Overall survival (OS) is the duration from date of randomization to date of death from any cause. Participants were censored at the date they were last known to be alive.
Time Frame: Baseline to date of death from any cause (up to 37.06 months)
Population: All randomized participants with FR-α Cytoplasm or Membrane H scores. Participants censored: FR-α Positive Cytoplasm n=21, 15 and Negative n=4, 3; FR-α Membrane Positive n=16, 8 and Negative n=9, 10 for Pem/Carbo/Bev and Pac/Carbo/Bev arms, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Number analyzed (Participants) | 98 | 82
months
  FR-α Cytoplasm Positive (H score > 0; n=64, 53) | 14.4 [11.4 to 22.2] | 14.3 [11.2 to 18.2]
  FR-α Cytoplasm Negative (H score = 0; n=34, 29) | 12.0 [9.6 to 16.9] | 11.2 [5.7 to 14.4]
  FR-α Membrane Positive (H score > 0; n=39, 22) | 19.2 [10.5 to 30.8] | 15.5 [11.2 to NA] — Not calculable due to the low number of participants reaching endpoint event of death.
  FR-α Membrane Negative (H score = 0; n=59, 60) | 12.9 [9.6 to 16.7] | 11.3 [8.8 to 14.7]
Statistical Analysis 1: Comparison: Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.891, Regression, Cox — p-value for FR-α Cytoplasm Positive (H score > 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.970, 95% CI 2-sided [0.622 to 1.511]
Statistical Analysis 2: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.060, Regression, Cox — p-value for FR-α Cytoplasm Negative (H score = 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.592, 95% CI 2-sided [0.342 to 1.023]
Statistical Analysis 3: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.905, Regression, Cox — p-value for FR-α Membrane Positive (H score > 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.960, 95% CI 2-sided [0.490 to 1.880]
Statistical Analysis 4: Comparison: Pem/Carbo/Bev vs Pac/Carbo/Bev; Test type: Superiority or Other; p = 0.455, Regression, Cox — p-value for FR-α Membrane Negative (H score = 0) comparing treatment arms and was not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.859, 95% CI 2-sided [0.575 to 1.281]

ADVERSE EVENTS:
Description: Deaths due to progressive disease are not considered adverse events and reported in the participant flow. All randomized participants who received at least 1 dose of study drug during the specified treatment phase.
Groups:
- Pem/Carbo/Bev: Induction:
  Bevacizumab: Induction therapy 15 milligrams per kilogram (mg/kg) intravenously (IV) every 21 days for up to 4 cycles of 21 days Pemetrexed: Induction therapy 500 milligram per meter squared (mg/m^2) IV every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days Carboplatin: Induction therapy of 6 area under the concentration curve (AUC 6) IV every 21 days for up to 4 cycles of 21 days
  Maintenance:
  Pemetrexed: Maintenance therapy 500 mg/m^2 IV every 21 days (with bevacizumab) until progressive disease or treatment discontinuation Bevacizumab: Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.
- Pac/Carbo/Bev: Induction:
  Paclitaxel: Induction therapy 200 milligram per meter squared (mg/m ²) intravenously (IV) every 21 days (with carboplatin and bevacizumab) for up to 4 cycles of 21 days Bevacizumab: Induction therapy 15 mg/kg IV every 21 days for up to 4 cycles of 21 days Carboplatin: Induction therapy 6 area under the concentration curve (AUC 6) IV every 21 days for up to 4 cycles of 21 days
  Maintenance:
  Bevacizumab: Maintenance therapy 15 mg/kg IV every 21 days until progressive disease or treatment discontinuation.
Arm/Group | Pem/Carbo/Bev | Pac/Carbo/Bev
Serious Adverse Events (participants affected / at risk) | 188/442 | 181/443
Other Adverse Events (participants affected / at risk) | 430/442 | 433/443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pem/Carbo/Bev (N=442) | Pac/Carbo/Bev (N=443)
Anaemia (Blood and lymphatic system disorders) | 18 (50) | 5 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7) | 13 (13)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (7) | 0 (0)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 10 (15) | 9 (9)
Pancytopenia (Blood and lymphatic system disorders) | 3 (5) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (20) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (4)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (4) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 3 (3)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (4) | 1 (2)
Myocardial infarction (Cardiac disorders) | 6 (6) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (8)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2 (3) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (9) | 7 (9)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (6)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (4) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 5 (5)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (4)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 2 (7) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (17) | 11 (21)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (4) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (20) | 11 (12)
Asthenia (General disorders) | 2 (4) | 9 (15)
Chest pain (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 1 (1) | 2 (2)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (4) | 3 (5)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (7)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 2 (3) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (6) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 4 (5)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (3)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (3)
Cellulitis (Infections and infestations) | 3 (5) | 3 (3)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 3 (8)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Hepatitis c (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Infectious peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (7) | 0 (0)
Meningitis herpes (Infections and infestations) | 0 (0) | 1 (2)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (10) | 1 (2)
Pneumonia (Infections and infestations) | 28 (39) | 27 (42)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (17)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (7) | 2 (2)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (3) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (14)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (15) | 1 (2)
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspiration pleural cavity (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 20 (27) | 21 (26)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 8 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Starvation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (8) | 4 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (6) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (8)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/235 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (3)
Cerebral ischaemia (Nervous system disorders) | 1 (2) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 5 (9) | 3 (4)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (7)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (3)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (11)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 2 (2)
Unresponsive to stimuli (Nervous system disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 5 (5) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (2)
Mental status changes (Psychiatric disorders) | 4 (4) | 2 (3)
Nephrotic syndrome (Renal and urinary disorders) | 1 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (7) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 7 (10) | 4 (5)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (30) | 2 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (14) | 8 (18)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 3 (6)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 6 (9)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (21) | 9 (14)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 4 (4)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (16) | 14 (34)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (5) | 1 (7)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 3 (5)
Intra-abdominal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (5) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pem/Carbo/Bev (N=442) | Pac/Carbo/Bev (N=443)
Anaemia (Blood and lymphatic system disorders) | 177 (1367) | 136 (793)
Leukopenia (Blood and lymphatic system disorders) | 73 (387) | 76 (362)
Neutropenia (Blood and lymphatic system disorders) | 170 (733) | 219 (790)
Thrombocytopenia (Blood and lymphatic system disorders) | 159 (829) | 105 (452)
Lacrimation increased (Eye disorders) | 31 (405) | 2 (12)
Abdominal pain (Gastrointestinal disorders) | 42 (171) | 39 (113)
Constipation (Gastrointestinal disorders) | 181 (1380) | 166 (931)
Diarrhoea (Gastrointestinal disorders) | 100 (536) | 118 (338)
Dyspepsia (Gastrointestinal disorders) | 49 (419) | 30 (155)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 25 (249) | 22 (178)
Nausea (Gastrointestinal disorders) | 236 (1465) | 223 (1157)
Stomatitis (Gastrointestinal disorders) | 61 (321) | 44 (159)
Vomiting (Gastrointestinal disorders) | 114 (369) | 108 (310)
Asthenia (General disorders) | 40 (230) | 29 (178)
Fatigue (General disorders) | 268 (2793) | 257 (2273)
Mucosal inflammation (General disorders) | 51 (229) | 35 (110)
Oedema peripheral (General disorders) | 66 (466) | 40 (249)
Pain (General disorders) | 22 (87) | 31 (196)
Pyrexia (General disorders) | 35 (104) | 42 (57)
Sinusitis (Infections and infestations) | 33 (111) | 19 (53)
Upper respiratory tract infection (Infections and infestations) | 32 (103) | 26 (53)
Urinary tract infection (Infections and infestations) | 32 (84) | 42 (108)
Alanine aminotransferase increased (Investigations) | 37 (291) | 12 (47)
Aspartate aminotransferase increased (Investigations) | 33 (207) | 17 (52)
Blood creatinine increased (Investigations) | 25 (163) | 13 (29)
Haemoglobin decreased (Investigations) | 39 (322) | 22 (102)
Platelet count decreased (Investigations) | 29 (106) | 14 (39)
Weight decreased (Investigations) | 77 (464) | 68 (470)
Decreased appetite (Metabolism and nutrition disorders) | 133 (865) | 145 (912)
Dehydration (Metabolism and nutrition disorders) | 68 (194) | 54 (155)
Hyperglycaemia (Metabolism and nutrition disorders) | 38 (251) | 45 (236)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (70) | 33 (76)
Hypomagnesaemia (Metabolism and nutrition disorders) | 34 (169) | 30 (186)
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 (272) | 107 (967)
Back pain (Musculoskeletal and connective tissue disorders) | 60 (299) | 64 (441)
Bone pain (Musculoskeletal and connective tissue disorders) | 16 (83) | 33 (204)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 33 (197) | 21 (141)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 42 (273) | 31 (246)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (150) | 60 (394)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (200) | 44 (413)
Dizziness (Nervous system disorders) | 77 (404) | 63 (298)
Dysgeusia (Nervous system disorders) | 67 (551) | 47 (283)
Headache (Nervous system disorders) | 82 (516) | 67 (343)
Neuropathy peripheral (Nervous system disorders) | 42 (413) | 145 (1394)
Paraesthesia (Nervous system disorders) | 11 (85) | 24 (255)
Peripheral sensory neuropathy (Nervous system disorders) | 19 (218) | 73 (888)
Anxiety (Psychiatric disorders) | 52 (407) | 44 (379)
Confusional state (Psychiatric disorders) | 19 (95) | 23 (48)
Depression (Psychiatric disorders) | 52 (402) | 47 (414)
Insomnia (Psychiatric disorders) | 69 (535) | 87 (719)
Proteinuria (Renal and urinary disorders) | 63 (435) | 54 (449)
Cough (Respiratory, thoracic and mediastinal disorders) | 91 (549) | 86 (568)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 32 (257) | 17 (126)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 88 (558) | 85 (503)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 117 (800) | 98 (599)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 41 (140) | 33 (115)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 29 (205) | 19 (153)
Alopecia (Skin and subcutaneous tissue disorders) | 34 (445) | 193 (2024)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (72) | 30 (91)
Rash (Skin and subcutaneous tissue disorders) | 42 (239) | 56 (177)
Hypertension (Vascular disorders) | 74 (800) | 70 (678)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days